CLINICAL TRIAL: NCT00019734
Title: Immunization of Patients With Metastatic Melanoma Using Recombinant Fowlpox and Vaccinia Viruses Encoding the Tyrosinase Antigen
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067075; NCI-99-C-0095; NCI-T99-0025; NCT00001811 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-05-28 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2007-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: fowlpox virus vaccine vector
Biological: vaccinia-tyrosinase vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of vaccine therapy with and without interleukin-2 in treating patients who have metastatic melanoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine efficacy of recombinant fowlpox and vaccinia viruses encoding tyrosinase antigen, administered with or without low-dose interleukin-2 (IL-2), in terms of response, in patients with metastatic melanoma.
* Compare the response rate in patients to this vaccination administered with high-dose IL-2 to that in similar patients on previous trials treated with high-dose IL-2 alone.
* Determine the immunological response in patients treated with this regimen.

OUTLINE: This is a randomized study. Patients are randomized to one of three treatment arms.

* Arm I: Patients receive recombinant fowlpox vaccine IM on day 1 followed 4 weeks later by recombinant vaccinia vaccine IM. Treatment repeats for a minimum of 4 vaccinations.
* Arm II: Patients receive vaccinations as in arm I plus low-dose interleukin-2 (IL-2) subcutaneously daily on days 2-13 after each vaccination.
* Arm III: Patients receive vaccinations as in arm I plus high-dose IL-2 IV over 15 minutes every 8 hours on days 2-5 after each vaccination.

Patients with stable disease or a minor, mixed, or partial response after four immunizations (1 course) may receive a second course of the same regimen beginning 4-6 weeks after the first course. After the second course, patients with tumor regression may continue to receive treatment in the absence of unacceptable toxicity until best response is achieved.

Patients are followed at 4-6 weeks.

PROJECTED ACCRUAL: A total of 73 patients (13-20 for arm I, 13-20 for arm II, and 19-33 for arm III) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma that has failed standard treatment
* No ocular or mucosal melanoma as primary site
* Measurable disease
* No existing brain metastases

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0 or 1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 90,000/mm3
* No coagulation disorder

Hepatic:

* Bilirubin no greater than 1.6 mg/dL
* AST/ALT less than 3 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 1.6 mg/dL

Cardiovascular:

* No major cardiovascular illness

Pulmonary:

* No major respiratory illness

Immunologic:

* HIV negative
* No autoimmune disease
* No primary or secondary immunodeficiency
* No allergy to eggs
* No history of allergy or untoward reaction to prior smallpox vaccination

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to avoid close contact with children under 5 years, pregnant women, people with active or a past history of eczema or other eczematoid skin disorders, and immunosuppressed people for at least 2 weeks after each vaccinia virus vaccination
* No active systemic infections
* No active atopic dermatitis or active or past history of eczema
* No concurrent active extensive psoriasis, severe acneiform rash, impetigo, varicella zoster, burns, or other traumatic or pruritic skin conditions or open wounds
* Surgical scars must be healed
* Healed surgical stomas (e.g., colostomy) allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior recombinant vaccinia or fowlpox vaccines for melanoma
* At least 3 weeks since prior systemic biologic therapy for melanoma

Chemotherapy:

* At least 3 weeks since prior systemic chemotherapy for melanoma

Endocrine therapy:

* At least 3 weeks since prior systemic endocrine therapy for melanoma
* No concurrent steroid therapy

Radiotherapy:

* At least 3 weeks since prior systemic radiotherapy for melanoma

Surgery:

* Prior surgery allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne L. Topalian, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States